CLINICAL TRIAL: NCT05414006
Title: Effect of S-ketamine in Cesarean Section Combined Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: S-ketamine and CS hyperalgesia
Record Dates: First submitted 2022-06-01; First posted 2022-06-10 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Pain
Keywords: S-ketamine; Cesarean Section; hyperalgesia
MeSH Terms: conditions — Pain, Postoperative; Hyperalgesia | interventions — Esketamine; Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: According to different groups, s-ketamine and placebo were given respectively According to the different PCA methods, different subgroups were included
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group E1 (Experimental): S-ketamine was administered intravenously after delivery，patient controlled epidural analgesia（PCEA）was administered postoperatively PCEA formula：（10μg/ml hydromorphone+0.11% ropivacaine) 200ml
  Interventions: Drug: S-ketamine
- Group E2 (Experimental): S-ketamine was administered intravenously after delivery，patient controlled intravenous analgesia（PCIA) was administered postoperatively PCIA formula：（100μg/ml hydromorphone) 100ml
  Interventions: Drug: S-ketamine
- Group C1 (Placebo Comparator): placebo was administered intravenously after delivery，patient controlled epidural analgesia（PCEA) was administered postoperatively PCEA formula：（10μg/ml hydromorphone+0.11% ropivacaine) 200ml
  Interventions: Drug: S-ketamine
- Group C2 (Placebo Comparator): placebo was administered intravenously after delivery，patient controlled intravenous analgesia（PCIA） was administered postoperatively PCIA formula：（100μg/ml hydromorphone) 100ml
  Interventions: Drug: S-ketamine

INTERVENTIONS:
Drug: S-ketamine — S-ketamine or placebo were given to the fetus after delivery Patient-controlled intravenous analgesia or patient-controlled epidural analgesia were administered postoperatively
  Other Names: Patient controlled analgesia

SUMMARY:
To compare the anti-hyperalgesia effect between S-ketamine with placebo for Maternal receiving elective Cesarean Section under Combined spinal and epidural analgesia.

Based on this study the investigators intend to verify the role and potential mechanism of S-ketamine combined anesthesia in alleviating hyperalgesia after cesarean section, prove that it can reduce hyperalgesia and postoperative pain. explore the role of S-ketamine in alleviating postoperative hyperalgesia in different PCA ways and explore the safety of S-ketamine in the perilactation

ELIGIBILITY:
Inclusion Criteria:

* ASA status I-III
* Age 20 to 45
* 37-42 weeks gestation
* undergo elective cesarean section with subarachnoid anesthesia
* participate in this study and sign informed consent

Exclusion Criteria:

* Patients with contraindications for cesarean section
* Patients with contraindications of combined spinal and epidural anesthesia
* Patients with severe systemic disease
* Alcoholism and long-term use of anti-inflammatory and analgesic drugs
* Patients who were unable to cooperate or refused to participate in the trial
* Patients with contraindications to esketamine and hydromorphone

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Maximum pain score (NRS socre) at 0-24 hours postoperatively | From ending of the surgery to 24 hours postoperatively
  NRS score: Pain was assessed on a scale of 0-10, with 0 being no pain and 10 being most painful
Pain score (NRS socre) at 0-6 hours postoperatively | From ending of the surgery to 6 hours postoperatively
  NRS score: Pain was assessed on a scale of 0-10, with 0 being no pain and 10 being most painful
Pain score (NRS socre) at 6-12 hours postoperatively | From 6 hours postoperatively to 12 hours postoperatively
  NRS score: Pain was assessed on a scale of 0-10, with 0 being no pain and 10 being most painful
Pain score (NRS socre) at 12-24 hours postoperatively | From 12 hours postoperatively to 24 hours postoperatively
  NRS score: Pain was assessed on a scale of 0-10, with 0 being no pain and 10 being most painful

SECONDARY OUTCOMES:
The number of patient controlled analgesia pump pressed | 0-48 hours postoperatively
  When the patients felt pain, the patient controlled analgesia pump can be pressed once
Patient controlled analgesia pump analgesic consumption | 0-48 hours postoperatively
  The amount of the analgesic consumption
Pressure pain threshold at 30min after surgery | Change from baseline to 30 minutes postoperatively
  Pressure pain threshold was measured using pressure manometer in the forearm of dominant hand reported by kg/cm2
Pressure pain threshold at 24 hours after surgery | Change from baseline to 30 min postoperatively
  Pressure pain threshold was measured using pressure manometer in the forearm of dominant hand reported by kg/cm2
Pressure pain tolerance at 30min hours after surgery | Change from baseline to 24 hours postoperatively
  Pressure pain tolerance was measured using pressure manometer in the forearm of dominant hand reported by kg/cm2

CONTACTS AND LOCATIONS:
Overall Officials: HUANG HE, MD, Study Director — Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within five years

REFERENCES:
- [Derived] Zhang J, Sun D, Wang J, Chen J, Chen Y, Shu B, Huang H, Duan G. Exploring the Analgesic Efficacy and mechanisms of low-dose esketamine in pregnant women undergoing cesarean section: A randomized controlled trial. Heliyon. 2024 Jul 30;10(15):e35434. doi: 10.1016/j.heliyon.2024.e35434. eCollection 2024 Aug 15. PMID 39170110